CLINICAL TRIAL: NCT05685407
Title: Examining Caffeine as a Treatment for Antidepressant-induced Arousal Dysfunction in Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 00002778
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Female Sexual Arousal Disorder
Keywords: female sexual dysfunction; female sexual arousal disorder; caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caffeine (Experimental): During one of two counterbalanced experimental sessions, participants will ingest 300mg of caffeine orally via capsules.
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): During one of two counterbalanced experimental sessions, participants will ingest placebo orally via capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Caffeine — 300mg caffeine will be administered orally via capsules to participants with female sexual arousal disorder.
  Arms: Caffeine
Other: Placebo — A placebo pill that matches in size, shape, and color will be administered to participants with female sexual arousal disorder.
  Arms: Placebo

SUMMARY:
Antidepressants have negative effects on genital arousal function that hinder quality of life and jeopardize medication adherence. Moderate sympathetic nervous system (SNS) activation through exercise has shown promising results for improving antidepressant-induced genital arousal dysfunction. It is feasible that caffeine - an SNS stimulant - could improve antidepressant-induced genital arousal difficulties if ingested prior to sex. The goal of the present pilot study is to examine whether the acute administration of 300mg of caffeine increases genital arousal in women experiencing antidepressant-induced genital arousal difficulties. Women will attend two counterbalanced sessions in which they ingest either 300mg caffeine or placebo. Fifteen minutes after ingestion, they will view an erotic film while their heart rate and genital sexual arousal are measured. Caffeine could serve as a low-cost, widely accessible intervention with minimal side effects if efficacy is shown.

ELIGIBILITY:
Inclusion Criteria:

* Between the of ages 18-55
* Fluent in English
* Experience antidepressant-induced arousal difficulties
* Experience regular menstrual periods (i.e., not perimenopausal or menopausal)

Exclusion Criteria:

* A history or current diagnosis of panic attacks or panic disorder
* A history or current diagnosis of sexually transmitted disease(s)
* A history of major pelvic surgery that caused nerve damage
* Currently taking beta blockers, antipsychotics, anti-anxiolytics, hormonal contraceptives (unless the participant has been taking it for over 3 months), or any other medical treatment to enhance sexual response
* Other medical conditions or procedures that would preclude the participant's participation in the study (e.g., urinary tract infection, neurological impairment due to diabetes or stroke, or spinal cord damage)
* A history of childhood sexual abuse (CSA) that occurred prior to age 16

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Vaginal pulse amplitude via vaginal photoplethysmography | 15 minutes post-ingestion of caffeine and placebo
  Vaginal pulse amplitude reflects phasic changes in vaginal engorgement with each heart beat, where higher amplitudes indicate higher levels of blood flow

SECONDARY OUTCOMES:
Subjective sexual arousal via Heiman and Rowland's (1983) Film Scale | 30 minutes post-ingestion of caffeine and placebo
  Discrete measurement of the construct was calculated by summing the scores of the three original subjective sexual arousal items from Heiman and Rowland's (1983) Film Scale, which assesses sexual arousal as well as positive and negative affect in response to an erotic film. These three items include an assessment of overall "sexual arousal," a sense of "mental sexual arousal," and one reverse-scored item on feeling "sexually turned off." On two occasions during the experiment (immediately following the first neutral-erotic film sequence and immediately following the second neutral-erotic film sequence), participants rated the degree to which they experienced each of the three items on a 7-point Likert scale (where higher scores indicate higher subjective sexual arousal), and then the three scores were combined into a single subjective sexual arousal score for each of the two time points.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy M Meston, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Sexual Psychophysiology Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT05685407/Prot_ICF_000.pdf